CLINICAL TRIAL: NCT03712176
Title: Descriptive Observational Study of the Evolution of the Lifestyle Alteration in Patients With Breast Cancer
Acronym: SPENCER
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0310
Record Dates: First submitted 2018-07-20; First posted 2018-10-19 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 : chemotherapy and radiotherapy: 50 women aged between 18 and 65 with first non-metastatic breast cancer treated by surgery and adjuvant therapy (chemotherapy and radiotherapy)
  Interventions: Behavioral: Lifestyle alteration
- Cohort 2 : radiotherapy only: 150 women aged between 18 and 65 with first non-metastatic breast cancer treated with surgery and adjuvant therapy (radiotherapy only).
  Interventions: Behavioral: Lifestyle alteration

INTERVENTIONS:
Behavioral: Lifestyle alteration — Patients will receive self-report questionnaires to evaluate their quality of life, fatigue level, anxiety and depression, cognitive complaint, cognitive efficiency, nutritional quality and food preferences, and sedentary behavior. Patients will also do tests to determine their physical conditions : six-minute walk test (6MWT), 30-s chair-stand test. The intervention will be done at three stages of the patient's care pathway: 1 / before the adjuvant surgery (baseline), 2 / at 6 months after the surgery and chemotherapy 3 / at 7 months after radiotherapy treatment.

SUMMARY:
Scientific context: With more than one million cases per year, breast cancer is the most common female cancer. All treatments such as surgery, chemotherapy, radiotherapy or hormone therapy lead to major changes patients' lifestyle. These treatments can lead to a decrease of physical activity due to fatigue and also changes in the diet. Sometimes, chemotherapy induces nutritional aversions and can cause weight gain that is known to increase the risk of recurrence. Cognitive complaints are also frequent, in particular in patients who received chemotherapy and can also lead to quality of life's alteration

Fatigue assessed with prevalence between 70 % and 100 % is usually a part of a series of symptoms including anxiety, depression, pain, sleep disturbance, decreased activity level, nutritional changes and pre-existent comorbidities. These symptoms can lead to an alteration of the quality of life. The chemotherapy involves disturbances at physiological, psychological and social levels and eating disorders leading to changes in eating habits which can lead to weight loss or weight gain. To limit these deleterious changes in lifestyle, increased physical activity, specialized counseling and nutritional monitoring may be recommended.

According to current knowledge there is no prospective study that evaluated different lifestyle changes according to different types of patients and the appearance of the installation of these symptoms during the patient pathway.

Research hypothesis: the study hypothesis is that description of the evolution of the quality of life and, physical, nutritional and cognitive parameters in a population of patients with non-metastatic breast cancer will better characterize these patients in order to propose an appropriate and personalized rehabilitation intervention.The investigators propose this feasibility study consisting of 2 cohorts of patients according to the adjuvant therapy given (+/- chemotherapy) after the primary breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 65 years old
* Breast invasive or in situ cancer (all histology), unilocal or multilocal tumor
* Treatment by first surgery and adjuvant radiotherapy validated at the multidisciplinary consultation meeting with +/- adjuvant chemotherapy (all chemotherapy)
* Patient reading and understanding the French language
* Non-opposition of patient

Exclusion Criteria:

* Patient with a history of treated breast cancer
* Presence of metastasis
* Other cancer or severe disease under evaluation or treatment at baseline (to avoid selection bias)
* Patient with psychiatric disorders
* Patient under protection status
* Pregnant or nursing women or absence of contraception in a patient of childbearing age

Withdrawal Criteria :

- Other cancer or severe illness diagnosed during the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women between 18 and 65 years old with first non-metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
The evolution of the quality of life | Cohorte 1 : at 7 months after radiotherapy treatment / Cohorte 2 : at 10 weeks after radiotherapy treatment
  The evolution of the quality of life will be evaluated by the FACT-B questionnaire (Functional Assessment of Breast Cancer Therapy). The FACT-B is a 37-item questionnaire divided into five subscales namely physical, social/family, emotional, functional well-beings, and the additional concerns for breast cancer. Each item is rated on a 5-point Likert scale. The FACT-B total score is the sum of scores of all five subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie JACQUIN-COURTOIS, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hôpital Henry Gabrielle, Saint-Genis-Laval, France